CLINICAL TRIAL: NCT02477033
Title: A Placebo-controlled Cross-over Randomized Study to Investigate the Impact of Butyricicoccus Pullicaecorum in Healthy Human Volunteers
Brief Title: Impact of Butyricicoccus Pullicaecorum in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Professor Kristin Verbeke, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ML9449
Record Dates: First submitted 2015-06-12; First posted 2015-06-22 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Butyricicoccus pullicaecorum (Active Comparator): Lyophilized Butyricicoccus pullicaecorum 25-3T bacteria, encapsulated with a pH-resistent coating.
  Interventions: Dietary Supplement: Butyricicoccus pullicaecorum 25-3T
- Placebo (maltodextrin) (Placebo Comparator): Lyophilized maltodextrin, encapsulated with a pH-resistent coating.
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Butyricicoccus pullicaecorum 25-3T
  Other Names: LMG 24109T; CCUG 55265T
  Arms: Butyricicoccus pullicaecorum
Other: Maltodextrin
  Arms: Placebo (maltodextrin)

SUMMARY:
During this project the safety, tolerability and effect on gut microbiota of oral administration of Butyricicoccus pullicaecorum was investigated in healthy human volunteers by a placebo-controlled cross-over randomized study.

DETAILED DESCRIPTION:
Intervention periods were 4 weeks, with daily intake of 1 capsule. Wash-out periods were 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 28 kg/m²
* Good general health
* Regular eating pattern (3 meals/day on at least 5 days/week)

Exclusion Criteria:

* Chronic gastrointestinal disease (Crohn's disease, ulcerative colitis, irritable bowel syndrome, chronic constipation or chronic diarrhea)
* Surgery of the gastrointestinal tract (except for an appendectomy)
* Use of antibiotics during the month preceding the study
* Use of medication or dietary supplements influencing gut transit or intestinal microbiota during the month preceding the study. Examples of such medication/dietary supplements are antispasmodics (e.g. buscopan), antidiarrheal medication (e.g. imodium), probiotic medication (e.g. lacteol, enterol)
* Intake of pre- or probiotics during the study or during the month preceding the study
* Being on a weight-loss diet during the study or during the month preceding the study
* Extreme dietary habits (e.g. vegan, Atkins diet, Montignac diet)
* Females who are pregnant, lactating or planning to become pregnant during the study period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Safety profile of Butyricicoccus pullicaecorum intake (composite outcome measure), measured by abdominal complaints surveys, standard blood tests and fecal calprotectin measurements | 1 year

SECONDARY OUTCOMES:
The effect of Butyricicoccus pullicaecorum intake on gut microbiota composition, measured by 16S rDNA Illumina profiling of the bacterial communities | 1 year
The effect of Butyricicoccus pullicaecorum intake on gut microbiota activity, measured by GC-MS analysis of the fecal volatile organic compounds | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- KULeuven, Leuven, Vlaams-Brabant, Belgium